CLINICAL TRIAL: NCT06808971
Title: A Phase II Clinical Trial of Adebrelimab Combined With Nab-paclitaxel, Oxaliplatin and Tegafur Gimeracil Oteracil Potassium Capsule for Perioperative Treatment of Locally Advanced Resectable Gastric/Gastroesophageal Adenocarcinoma
Brief Title: Adebrelimab Combined With Nab-paclitaxel, Oxaliplatin and Tegafur (AOS) for Perioperative Treatment of Locally Advanced Resectable GC/GEJ
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LIN YANG, Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5105
Record Dates: First submitted 2025-01-25; First posted 2025-02-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-01

CONDITIONS: Gastric Adenocarcinoma; Gastro-esophageal Junction Adenocarcinoma
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab, Nab-paclitaxel, Oxaliplatin, Tegafur Gimeracil Oteracil Potassium Capsule (Experimental): Adebrelimab combined with Nab-paclitaxel, Oxaliplatin and Tegafur Gimeracil Oteracil Potassium Capsule
  Interventions: Drug: Adebrelimab, Nab-paclitaxel, Oxaliplatin, Tegafur Gimeracil Oteracil Potassium Capsule

INTERVENTIONS:
Drug: Adebrelimab, Nab-paclitaxel, Oxaliplatin, Tegafur Gimeracil Oteracil Potassium Capsule — Adebrelimab combined with Nab-paclitaxel, Oxaliplatin andTegafur Gimeracil Oteracil Potassium Capsule

SUMMARY:
This study is a single-arm, prospective, phase II clinical trial. The patients are diagnosed with resectable locally advanced (cT3-4N+M0) gastric adenocarcinoma and esophageal gastric adenocarcinoma that had not been treated before.

After signing the informed consent form, patients will be screened for the study treatment of Adebrelimab combined with AOS. After 2 cycles of treatment, MDT assessments before surgery will be carried out. Patients with no disease progression will receive one more cycle of treatment before surgery. For patients who have undergone radical surgery, they will continue to receive 3 cycles of the immunochemotherapy after the operation (a total of 6 cycles of combined treatment before and after surgery), followed by Adebrelimab single treatment for up to a year (16 cycles).

Patients whose disease progressed that can not be surgically removed after preoperative treatment will be treated by the oncology physicians according to clinical routines.

DETAILED DESCRIPTION:
This study is a single-arm, single-center, prospective, phase II clinical trial. The study subjects are patients with resectable locally advanced (cT3-4N+M0) gastric adenocarcinoma and esophageal gastric adenocarcinoma that had not been treated before.

A team of doctors, which includes the oncology physicians, surgeons and radiologists, will be in charge of the response assessment every two cycles of the study treatment. Then they will together decide whether the patient can receive radical surgery.

After signing the informed consent form, patients will be screened for the study treatment of Adebrelimab combined with AOS. After 2 cycles of treatment, MDT assessments before surgery will be carried out. Patients with no disease progression will receive one more cycle of treatment before surgery. For patients who have undergone radical surgery, they will continue to receive 3 cycles of the immunochemotherapy after the operation (a total of 6 cycles of combined treatment before and after surgery), followed by Adebrelimab single treatment for up to a year (16 cycles).

Patients whose disease progressed that can not be surgically removed after preoperative treatment will be treated by the oncology physicians according to clinical routines.

Safety follow-up: D1 per treatment cycle, before surgery, 30 days after the last study treatment.

Disease progression follow-up: every 2 treatment cycles (6 weeks) before the surgery. Every 3 months after the surgery for 2 years. Every 6 months after the surgery for 2 to 5 years, and once a year after five years.

Survival follow-up: Since the last cycle of treatment, it is carried out every three months until the patient died, missed or withdrew from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study and sign informed consent forms;
2. 18-75 years old;
3. Patients whose tumor has been pathologically diagnosed as gastric adenocarcinoma or gastroesophageal junction adenocarcinoma, and has not received any type of antitumor treatment (such as surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.);
4. Confirmed TNM staging by CT or MRI as resectable cT3-4N+M0;
5. ECOG score is 0-1;
6. Patients who are able to swallow pills and capsules normally;
7. Patients whose expected survival period is longer than 12 weeks;
8. The function of important organs meets the following requirements:

A. Absolute number of neutrophils (ANC) ≥1.5×10^9/L B. Platelet number ≥90×10^9/L; C. Hemoglobin ≥90g/L; D.Total bilirubin ≤1.5×ULN; ALT, AST and/or AKP≤2.5×ULN; E. Serum creatinine ≤1.5×ULN or creatinine clearance rate >60mL/min (Cockcroft-Gault); F. Activated partial thromboplastin time (APTT) and international standardization ratio (INR) ≤1.5×ULN (for anticoagulation treatments using stable doses such as low-molecular heparin or warfarin and INR can be screened within the expected treatment range of anticoagulants); 9. Female patients with fertility must undergo a blood pregnancy test within 72 hours before the first administration of the drug and the result is negative. During the study period and at least 6 months after the last dose of the study drug, a medically approved contraceptive measure (such as intrauterine birth control device, contraceptive pill or condom) must be used; for men, it should be surgery, sterilization, or agree to use effective contraception during the study period and within 6 months after the last dose of the study drug.

Exclusion Criteria:

1. Patients who are known to have peritoneal metastasis or positive peritoneal lavage cytology (CY1P0) or have distant metastasis;
2. Patients whose tumor can not be resected by surgery for tumor reasons or comorbidity or patients who refuse to undergo surgery;
3. Patients who have other malignant tumors within the past 5 years or at the same time, except for cured skin basal cell carcinoma, cervical in situ and breast cancer in situ;
4. The toxicity of previous anti-tumor treatment has not recovered to CTCAE≤grade one (NCI CTCAEv5.0), except for hair loss (any level allowed) and peripheral neuropathy (need to be ≤grade two );
5. Active bleeding;
6. Patients who had gastrointestinal perforation, abdominal abscess or recent intestinal obstruction or imaging and clinical symptoms with intestinal obstruction in the past 3 months;
7. Uncontrollable hypertension, symptomatic cardiac insufficiency, and severe heart disease within 6 months, including but not limited to:

(1) Acute coronary syndrome; (2) Arrhythmias that require drug treatment or have clinical significance, or do not interrupt the use of drugs that may lead to QT prolongation during the research period; (3) Acute myocardial infarction; (4) Heart failure; (5) Any other heart disease judged by the researchers to be unsuitable for participating in this trial.

8. Patients who have active ulcers, unhealed wounds or fractures; 9. Patients who need antimicrobial treatment in the stage of active infection; 10. Active hepatitis (Hepatitis B reference: HBsAg positive and HBV DNA ≥500IU/ml; hepatitis C reference: HCV antibody positive and HCV virus copy number > normal value upper limit); 11. Patients with congenital or acquired immunodeficiency; 12. Patients who are planning to receive or have previously received organ or allogeneic bone marrow transplantation; 13. At present, patients who are accompanied by interstitial pneumonia or interstitial lung disease, or who have a previous history of interstitial pneumonia or interstitial lung disease that require hormone treatment, or other patients who may interfere with the judgment and treatment of immune-related pulmonary toxicity, fibrosis, organic pneumonia (such as occlusion bronchiolitis), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia, or screening CT showing active pneumonia or severe pulmonary function impairment; active pulmonary tuberculosis; 14. Patients with any active autoimmune diseases or a history of autoimmune diseases with the possibility of recurrence [including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism (patients who can only be controlled by hormone replacement therapy can be included in the group)]; patients with skin diseases that do not require systemic treatment, such as leukoplakia, psoriasis, hair loss, patients with type I diabetes that can be controlled by insulin treatment or have a history of asthma, but who have been completely relieved in childhood and do not require any intervention can be included in the group; asthma patients who need the intervention of bronchodilators cannot be included in the group; 15. Patients who are using immunosuppressive drugs or systemic corticosteroid treatment within 7 days before joining in the group to achieve the purpose of immunosuppression (>10mg/day of prednisone or other equivalent drugs); 16. Patients who have received live attenuated vaccine within 28 days before joining in the group, or need to inject such vaccines during treatment or within 60 days after the last dose; 17. Oral or intravenous antibiotics or intravenously within 4 weeks before joining the group (except for preventive antibiotics administered intravenously for no more than 48 hours); 18. Known allergies to any study drugs or excipients; 19. Participated in clinical research of other drugs 4 weeks before joining in the group; 20. Lactating women; 21. According to the researcher's judgment, the patient has other factors that may affect the research results or cause the forced termination of this study, such as alcoholism, drug abuse, other serious diseases (including mental illness that need combined treatment, and serious laboratory examination abnormalities, accompanied by family or social factors, which will affect the safety of patients);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate (pCR) | At the time of pathological diagnosis
  The percentage of patients who undergone surgery with tumor regression grade of class one, which there is no tumor cell residue in the tumor lesions.

SECONDARY OUTCOMES:
Event Free Survival (EFS) | From the time of the first study treatment to the first occurrence of any of the following events: disease progression, local or distant recurrence and metastasis, death, etc.
  From the beginning of the study treatment to the first occurrence of any of the following events: disease progression, local or distant recurrence and metastasis, death, etc.
major pathological response rate (MPR) | At the time of pathological diagnosis
  The percentage of patients with TRG grade two, which the tumor residues are rare in tumor lesions.
Treatment safety | Recording the adverse events occurs from the time of the first dose of study treatment to 30 days after the last medication.
  The adverse events occur during the study treatment, including that occurs during the immunochemotherapy and the surgery.

OTHER OUTCOMES:
biomarker | Baseline, two cycles of treatment before surgery, after surgery before adjuvant treatment, every three months during the study treatment, when disease progressed.
  PD-L1, TMB, ctDNA, plasma cytokine, plasma proteome

CONTACTS AND LOCATIONS:
Overall Officials: LIN YANG, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No